CLINICAL TRIAL: NCT02959957
Title: A Randomized, Controlled, Multicentre Trial of Collateral Damage on the Intestinal Microbiota Inferred by Temocillin Versus Cefotaxime in Patients Receiving Empirical Treatment for Febrile Urinary Tract Infections
Brief Title: Disturbance of the Intestinal Microbiota by Temocillin vs Cefotaxime in Treatment of Febrile Urinary Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Håkan Hanberger (Other Government)
Responsible Party: Sponsor-Investigator, Håkan Hanberger, Professor, Public Health Agency of Sweden
Organization: Public Health Agency of Sweden (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoHM/UVI 2015; 2015-003898-15 (EudraCT Number)
Record Dates: First submitted 2016-10-13; First posted 2016-11-09 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — temocillin; Cefotaxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temocillin (Experimental): Temocillin powder for solution för injection/infusion, per day 6 g (2 g three times per day). Treatment length 7-10 days of which at least 3 days administration with the study drug.
  Interventions: Drug: Temocillin
- Cefotaxime (Active Comparator): Cefotaxime powder for solution för injection/infusion, per day 3-6 g (1-2 g three times per day). Treatment length 7-10 days of which at least 3 days administration with the study drug.
  Interventions: Drug: Cefotaxime

INTERVENTIONS:
Drug: Temocillin — Total antibiotic treatment 7-10 days, of which at least 72 hours (9 doses) initial temocillin administration. In case of bacteraemia at baseline the total antibiotic treatment can be extended up to 14 days.
  Other Names: Negaban
  Arms: Temocillin
Drug: Cefotaxime — Total antibiotic treatment 7-10 days, of which at least 72 hours (9 doses) initial cefotaxime administration. In case of bacteraemia at baseline the total antibiotic treatment can be extended up to 14 days.
  Other Names: Claforan
  Arms: Cefotaxime

SUMMARY:
This study will evaluate the ecological impact on the intestinal microbiota and compare the safety and efficacy of temocillin compared to cefotaxime, in empiric treatment of febrile UTI. Half of participants will receive temocillin and the other half will receive cefotaxime.

DETAILED DESCRIPTION:
Temocillin is a narrow spectrum antibiotic with activity against gram negative bacteria inclusive many ESBL producing bacteria. Temocillin is approved and marketed in a few European countries since the 1980´s but not in Sweden.

The aim of the study is to find an ecological favorable alternative to cephalosporins in the treatment of this common indication.

The hypothesis is that treatment with temocillin causes less disturbances on the intestinal microbiota while at least comparable efficacy.

The study will be performed as an open prospective multicentre study with two parallel groups comparing 2 g temocillin three times daily with 1-2 g cefotaxim three times daily for 7-10 days in male and female adult patients with febrile urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age with suspected or confirmed febrile UTI, fulfilling at least one of the following signs and symptoms:

  * Flank pain or suprapubic pain, Tenderness over the kidney on physical examination, Urinary symptoms such as dysuria, urinary frequency or urinary urgency
* Fever ≥ 38.0°C (highest temperature recorded at home or at the hospital)
* Positive urinalysis tests (U-Nitrit and/or U-LPK)
* Have a pre-treatment baseline urinary culture obtained
* Require iv antibacterial treatment of the presumed infection
* Fertile women: Agree to practice highly effective anti-contraceptive methods from study-start to TOC
* Signed informed consent

Exclusion Criteria:

* Have a documented history of hypersensitivity or allergic reaction to any beta-lactam
* Pregnant or nursing women
* Receipt of any prior potentially therapeutic antibacterial agent within 1 month before randomisation and sampling for urine and faecal cultures. Exceptions will prior treatment with pivmecillinam or nitrofurantoin.
* Known chronic renal insufficiency (creatinine clearance < 10 mL/min at screening as estimated by Cockcroft-Gault), or receiving intermittent haemodialysis or peritoneal dialysis
* Known colonization with ESBL
* Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the subject or the quality of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with emergence of any of the two following events: Colonisation or infection with C. difficile and/or with Enterobacteriaceae resistant to 3rd generation cephalosporins. Measured in cultures from faecal samples. | Within 12 hours after the last dose of study drug.
  Superiority analysis.

SECONDARY OUTCOMES:
Number of patients with clinical cure in each treatment group. | 7-10 days after discontinuation of antibiotic treatment (parenteral and oral).
  Clinical cure defined as patient totally recovered with no remaining symptoms of UTI or no recurrence with symptoms or no need of further treatment against the current infection. Non-inferiority analysis.
Number of patients with early clinical response. | Within 12 hours after the 9th dose of study drug.
  Non-inferiority analysis.
Bacteriological cure per patient and per pathogen measured as negative urine Culture <1000 CFU/ml. | 7-10 days after discontinuation of antibiotic treatment (parenteral and oral).
  Non-inferiority analysis.
Early bacteriological response measured as negative urine Culture <1000 CFU/ml. | Within 12 hours after the 9th dose of study drug.
  Non-inferiority analysis.
Rate of patients with diarrhea (≥ 3 loose stools per day) | From the first dose of study drug until 7-10 days after discontinuation of antibiotic treatment (parenteral and oral).

OTHER OUTCOMES:
Frequency of adverse events | From the first dose of study drug until 4-6 weeks after discontinuation of antibiotic treatment (parenteral and per oral).

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Hanberger, Professor, Principal Investigator — University Hospital, Linkoeping
Locations (12):
- Sweden (12):
  - Karolinska University Hospital, Solna, Stockholm County
  - Helsingborg Hospital, Helsingborg
  - Centralsjukhuset Kristianstad, Kristianstad
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Vrinnevisjukhuset i Norrköping, Norrköping
  - Örebro University Hospital, Örebro
  - Östersund Hospital, Östersund
  - Capio S:t Görans hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - University Hospital of Umeå, Umeå
  - Västmanlands sjukhus i Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No